CLINICAL TRIAL: NCT06025318
Title: An Open-label, Balanced, Randomized, Two-period, Crossover, Single Dose Study to Compare the Bioavailability of PanCytoVir™ Oral Suspension (100mg/ml), in Healthy, Adult, Human Subjects Under Fed and Fasting Conditions
Brief Title: An Evaluation of the Effect of Food on the PK of a Novel PanCytoVir™ Suspension (100mg/ml), in Healthy, Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TrippBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VRS-23-001
Record Dates: First submitted 2023-08-24; First posted 2023-09-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Relative Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PanCytoVir™ 1000 mg fasted (Experimental): Single oral dose of PanCytoVir™ 1000 mg (100 mg/mL suspension) following an overnight fast
  Interventions: Drug: PanCytoVir™
- PanCytoVir™ 1000 mg fed (Experimental): Single oral dose of PanCytoVir™ 1000 mg (100 mg/mL suspension) following a standard, high-fat, high-calorie breakfast
  Interventions: Drug: PanCytoVir™

INTERVENTIONS:
Drug: PanCytoVir™ — PanCytoVir™ 100 mg/mL oral suspension

SUMMARY:
This is an open-label, balanced, randomized, two-period, crossover, single dose study to compare the relative bioavailability in normal healthy, adult, human subjects under Fed and Fasting conditions. Subjects will receive a single oral dose of probenecid oral suspension (100 mg/mL) under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy adult human subjects.
2. Subjects who are willing to participate and give informed consent
3. Subjects who are ≥ 18 years of age to ≤ 45 years of age and have a Body Mass Index between ≥18.5 to ≤ 30.0 kg/m2 extremes included, with weight of at least 50 kg.
4. Subjects with normal findings as determined by baseline history, physical examination and vital sign examination (blood pressure, pulse rate, respiration rate and body temperature).
5. Subjects with clinically acceptable findings as determined by haemogram, biochemistry, urine analysis, 12 lead ECG and chest X-ray.
6. Willingness to follow the protocol requirements especially abstaining from xanthine containing food or beverages (chocolates, tea, coffee or cola drinks) or grapefruit juice, any alcoholic products, the use of cigarettes and the use of tobacco products for 72.00 hours prior to dosing until after the last blood sample collection in each study period and adherence to food, fluid and posture restrictions.
7. No history of significant alcoholism.
8. Subject who have an estimated glomerular filtration rate (eGFR) value is >60ml/min.
9. Found negative in Alcohol test.
10. Found negative in urine test for drug abuse [Benzodiazepines, Barbiturates, Morphine, Cocaine, Amphetamines and Tetrahydrocannabinol (THC)].
11. Non-smokers, ex-smokers and moderate smokers will be included. "Moderate smokers are defined as someone smoking 10 cigarettes or less per day, ex-smokers are someone who completely stopped smoking for at least 3 months."

Exclusion Criteria:

1. History of allergic responses or hypersensitivity to Probenecid or other related drugs, or any of its ingredients.
2. Requiring medication for any ailment having enzyme-modifying activity in the previous 21 days, prior to dosing day.
3. Subjects who have taken prescription medications or over-the-counter products (including vitamins and minerals) within 14 days prior to administration of study drug
4. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
5. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, haematological, gastrointestinal, endocrine, immunological or psychiatric diseases.
6. Participation in a clinical drug study or bioequivalence study 90 days prior to period I dosing of the present study.
7. History of malignancy or other serious diseases.
8. Blood donation 90 days prior to period I dosing of the present study.
9. Subjects with positive HIV tests, HBsAg or Hepatitis-C tests.
10. History of problem in swallowing tablets/capsules/ Suspension.
11. Any contraindication to blood sampling.
12. Female subjects found positive serum (β) Beta- hCG (Human Chorionic Gonadotropin) test.
13. Lactating women (currently breast feeding).
14. Female subjects not confirming to using birth control measures, from the date of screening until the completion of the study. Abstinence, barrier methods (condom, diaphragm, etc.) are acceptable.
15. Use of hormonal contraceptives either oral or implants.
16. History of urinary retention, gastric retention and other severe decreased gastrointestinal motility conditions, uncontrolled narrow-angle glaucoma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
To assess food effect on PanCytoVir™ in healthy, adult, human subjects as assessed by Cmax | 7 days
  The drug concentration in plasma assessed by Cmax
To assess food effect on PanCytoVir™ in healthy, adult, human subjects as assessed by AUC | 7 days
  The drug concentration in plasma assessed by AUC

SECONDARY OUTCOMES:
the Incidence rates of AEs, TEAEs and Serious Adverse Events (SAEs) | 7 days
  Numbers and incidence rates of AEs, TEAEs and Serious Adverse Events (SAEs) will be tabulated using available version of Medical Dictionary for Regulatory Activities (MedDRA) preferred term (PT), system organ class (SOC), severity and relationship. A patient having the same AE will be counted only once in calculating frequency while patient having same AE with different start date then both will be considered for calculating frequency. If AE is with same start date but different criteria (severity, relationship to study medication and outcome), worst case/latest case (whichever applicable) will be considered. Incidence of AEs will be summarized with count (%).

CONTACTS AND LOCATIONS:
Overall Officials: David E Martin, PharmD, Study Director — TrippBio, Inc.
Locations (1):
- Vayam Research Solutions Limited, Gujarat, India, India

IPD SHARING:
Plan to Share IPD: No
Plans are currently being developed